CLINICAL TRIAL: NCT05823077
Title: Effects of Aromatherapy Massage in Menopausal Women With Knee Osteoarthritis: a Randomized Placebo-controlled Trial
Brief Title: Effects of Aromatherapy Massage in Menopausal Women With Knee Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: KTO Karatay University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KaratayUH8
Record Dates: First submitted 2023-04-08; First posted 2023-04-21 (Actual); Last update posted 2023-08-21 (Actual); Status verified 2023-04

CONDITIONS: Osteoarthritis, Knee
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — bergamot oil

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Bergamot (Experimental): In addition to 4 weeks of conventional treatment, Bergamot oil diluted with 1.5% sweet almond oil (4 drops of aromatic oil to 10 cc of sweet almond oil) will be used on the participants. After the oil is diluted, it will be heated up to 36oC. The participant will sit on the stretcher directly opposite the therapist, with the affected knee semi-flexed. The therapist will massage the affected knee for 15 minutes. After the massage, the knees will be wrapped with a towel for 5 minutes.
  Interventions: Other: Bergamot
- Placebo (Placebo Comparator): In addition to 4 weeks of conventional treatment, Pure sweet almond oil will be used for the participants. Sweet almond oil will be heated to 36oC. The participant will sit on the stretcher directly opposite the therapist, with the affected knee semi-flexed. The therapist will massage the affected knee for 15 minutes. After the massage, the knees will be wrapped with a towel for 5 minutes.
  Interventions: Other: Placebo
- Control (No Intervention): 4 weeks of conventional treatment.

INTERVENTIONS:
Other: Bergamot — The affected knee will be massaged with Bergamot oil for 4 weeks, 2 sessions per week.
  Arms: Bergamot
Other: Placebo — The affected knee will be massaged with sweet almond oil for 4 weeks, 2 sessions per week.
  Arms: Placebo

SUMMARY:
In this study, the effects of 4-week aromatherapy massage on pain, functionality, sleep quality and menopausal symptoms will be examined in individuals diagnosed with knee osteoarthritis during menopause.

DETAILED DESCRIPTION:
The aim of this study is to investigate the effect of aromatherapy massage performed with bergamot oil for 4 weeks on pain, function, sleep and menopausal symptoms in menopausal women with knee osteoarthritis. Participants will be randomly divided into 3 groups as Bergamot, placebo and control. In addition to the conventional treatment, the Bergamot group will receive 2 sessions of Bergamot oil per week for 4 weeks, and the placebo group will be massaged with 2 sessions of sweet almond oil for 4 weeks. the control group will continue conventional treatment for 4 weeks. All assessments will be performed before starting treatment and at the end of 4 weeks of treatment. Participants' pain will be evaluated by VAS, Functions by WOMAC, Sleep quality by PSQI, menopausal symptoms by Menopause Symptoms Evaluation scale. At the end of the study, the satisfaction of the participants will be evaluated with VAS.

ELIGIBILITY:
Inclusion Criteria:

* Being between the ages of 40-65,
* having entered the menopause,
* being diagnosed with knee OA,
* being at the level of OA 2-3,
* having pain at rest in the knee VAS ≥ 4.

Exclusion Criteria:

* Any knee surgery
* known allergies to the oils to be used

Ages: 40 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2023-05-24 (Actual); Primary Completion 2023-08-01 (Actual); Study Completion 2023-08-13 (Actual)

PRIMARY OUTCOMES:
Change from baseline in pain at 4 weeks | Baseline and 4 weeks
  The rest, activity and night pains of the participants will be evaluated with a 10 cm Visuak Analog Scale before the treatment and at the end of the 4-week application. "0" means no pain, "10" means excruciating pain. Results will be recorded in cm.

SECONDARY OUTCOMES:
Change from baseline in function at 4 weeks | Baseline and 4 weeks
  Participants' functions will be evaluated with Western Ontario and McMaster Universities Osteoarthritis Index. A minimum of "0" points and a maximum of "96" points can be obtained on the scale. High scores indicate high impairment and limitation of functional status and poor quality of daily life. Evaluations will be made before the study and after 4 weeks of practice.
Change from baseline in sleep quality at 4 weeks | Baseline and 4 weeks
  The sleep quality of the participants will be evaluated with Pittsburgh Sleep Quality Index . The total score is between 0-21. High scores indicate poor sleep quality. Evaluations will be made before the study and after 4 weeks of practice.
Change from baseline in menopause symphtoms at 4 weeks | Baseline and 4 weeks
  Participants' menopausal symptoms will be evaluated with the Menopause Symptoms Evaluation Scale. Higher scores indicate more menopausal symptoms. Evaluations will be made before the study and after 4 weeks of practice.
Patients satisfaction after the interventions | 4 weeks
  Participants' satisfaction with the treatment over pain and function will be evaluated with Visual Analog Scale. Higher score indicate more satisfaction. Evaluation will take place after 4 weeks of study.

CONTACTS AND LOCATIONS:
Locations (1):
- KTO Karatay University, Konya, Karatay, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided